CLINICAL TRIAL: NCT04056013
Title: Vicryl Rapide Versus Nonabsorbable Suture in Repair of Simple Traumatic Extremity and Trunk Lacerations in Adult Patients
Brief Title: Vicryl Rapide Versus Nonabsorbable Suture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Central California Faculty Medical Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019062
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Lacerations
Keywords: Traumatic lacerations; Vicryl Rapide; nonabsorbable suture; Suture

STUDY DESIGN:
Intervention Model Description: Patients meeting eligibility criteria will be randomized to treatment with either Vicryl Rapide or nonabsorbable suture. To ensure comparable numbers patients with buried sutures, there will also be 1 block of 8 patients that is randomized for absorbable or nonabsorbable closure in patients who are receiving buried sutures.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Absorbable (Active Comparator): Wound repaired with Vicryl Rapide absorbable suture
  Interventions: Device: Vicryl Rapide absorbable suture
- Nonabsorbable (No Intervention): Wound repaired with traditional nonabsorbable suture

INTERVENTIONS:
Device: Vicryl Rapide absorbable suture — In general, most laceration repair has been done with sutures on the surface of the skin that do not break down and fall off on their own, so after enough days have passed for the laceration to heal properly, the patient needs to return to the ED to have the sutures removed by cutting them off. These sutures are called "nonabsorbable". Some newer sutures have been designed to slowly dissolve on their own and fall out over several days. These are called "absorbable" sutures. You do not normally need to return to the ED for removal as these should slowly dissolve and fall out on their own.
  Arms: Absorbable

SUMMARY:
This will be a prospective, randomized controlled trial assessing noninferiority of Vicryl Rapide compared to nonabsorbable suture. The study will be conducted in the Community Regional Medical Center emergency department (ED). The aim of this study, then, is to prospectively determine if 3-month cosmesis for traumatic laceration repair of trunk/extremity lacerations in adult patients with Vicryl Rapide is noninferior to nonabsorbable suture.

DETAILED DESCRIPTION:
Study flyers will be posted in all doc boxes to ensure all ED personnel is aware of ongoing studies. Initial ED history and physical examination (standard procedure). Provider identifies patient who is felt to require suture closure. Provider will contact study staff that approved to consent patient to consent the patient for the study. After identification of a patient who meets inclusion criteria, the patient will be screened for exclusion criteria by the investigators using a preprinted form on the outside of the study envelope. If the patient has an exclusion criterion, this will be noted on this preprinted form and the form will be saved for further data analysis without any patient identifiers, and the patient will not be enrolled in the study. If the patient does not have exclusion criteria, the enrollment envelope will be opened and he/she will undergo the written consent process. After written consent is complete, the randomization envelope is opened. There will be a question asking if buried sutures will be needed as the group of patients needing buried sutures will have their own randomized packets to ensure a similar amount of buried suture patients are in both the Vicryl Rapide and nonabsorbable suture closure group. The study staff will then gather the following information regarding wound characteristics: Measure the length and width of the laceration, laceration location, presence of contamination, and if it is simple linear. The laceration will then be prepped for closure using whatever cleaning or anesthesia is felt to be appropriate by the practitioner. Suture closure will then occur with either Vicryl Rapide or nonabsorbable suture according to randomization direction in the envelope. After laceration closure, the practitioner will also write down on this paper the suture size and, for the nonabsorbable group, the type of suture used. The practitioner performing suture closure will also write down whether he/she is the nurse practitioner (NP), physician assistant (PA), emergency medicine (EM) faculty or EM resident. Patients will be given preprinted discharge instructions appropriate to whether Vicryl Rapide or nonabsorbable suture was used that gives information such as precautions for infection, information about how to do the 3-month follow-up, research coordinator contact information, and date to return for suture removal in the nonabsorbable group.

At 30 days post enrollment, the patient will receive a call from trained Institutional review board (IRB) approved study personnel. The pre-printed scripted form will ask questions to determine if the patient had any complications including infection, dehiscence, and, in the absorbable suture group, whether a return visit was needed to have the sutures removed.

At 30 days post enrollment, study personnel will also do a chart review collecting the following elements: Patient's age, ethnicity, gender, comorbid conditions including diabetes mellitus, renal insufficiency, liver disease, and immunodeficiency, ED vital signs, and whether patient was admitted or treated as outpatient for the index visit. The chart will also be reviewed examining for any revisit to the ED during those 30 days with any of the complications listed in the previous paragraph.

At three-months post enrollment, the research coordinator will work with the patient to arrange an appointment to take pictures of the wound. The patient will have their follow-up visit done at the Clinical Research Center at the University of California, San Francisco (UCSF) Fresno building. The photographs will be taken by study personnel with instructions on how to take these. At this time, the patient would be provided with a gift card and log book would be signed by the patient. The photographs are then prepared for submission to the plastic surgeon who will be evaluating them. Photographs will not have any patient identifiers other than a study number, and would be labeled with the anatomic area. The plastic surgeon, who is a blinded study staff to the study hypothesis, then assesses the cosmesis of the wound on a 100-mm visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-years or older

  * single laceration on trunk or extremity requiring suture closure
  * laceration length > 2-cm
  * wound to be closed with simple interrupted sutures

Exclusion Criteria:

* High infection potential
* Must have one of the following:

  * puncture wound

    * -highly contaminated
  * devitalized tissue requiring sharp debridement

    * -bite wounds
    * -> 24-hours-old

      * Low likelihood of good cosmesis
* Must have one of the following:

  -⁮dehisced wound from previous wound closure
  * -wound
  * -crush wound
  * -soft tissue deficit limiting complete apposition of wound edges
  * -significant overlying macerated/abraded tissue

    * Underlying tendon or cartilage involvement

      -⁮Wound greater than 10 cm in length
    * Significant wound healing problems
* Must have one of the following:

  * keloid formers
  * chronic steroid use
  * other: ______________________ ⁮-Inability to give written consent
* Must have one of the following:

  * non-English or non-Spanish speaker

    * altered mental status
  * incarcerated patient
  * No telephone number or unlikely to return for 3-month follow-up
* Must have one of the following:

  * homeless
  * psychiatric patient,
  * nursing home patient,
  * other: ______________________
  * More than one laceration needing suture repair on trunk or extremity (i.e. appropriate to proceed if second laceration is to face/neck)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
The two treatments will be compared by a noninferiority test | 3-Month
  For sample size determination, based on a previous study, we expected that the standard deviation (SD) for cosmesis scores would be 15 mm.10 With the minimum clinically important cosmetic difference of 12-mm, and assuming an alpha value of 0.05 and statistical power of 90%, we estimated that we would need 46 subjects in each group for a total of 96 patients (assuming a dropout rate of 40%), to detect this 12-mm difference in the groups' mean cosmesis scores.

SECONDARY OUTCOMES:
Percentage of patients needing further treatment | 30-days
  Follow-up call to determine if patient required further treatment beyond routine care

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chinnock, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Community Regional Medical Center, Fresno, California
  - Community Regional Trauma and Burn Center, Fresno, California

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Background] Karounis H, Gouin S, Eisman H, Chalut D, Pelletier H, Williams B. A randomized, controlled trial comparing long-term cosmetic outcomes of traumatic pediatric lacerations repaired with absorbable plain gut versus nonabsorbable nylon sutures. Acad Emerg Med. 2004 Jul;11(7):730-5. doi: 10.1197/j.aem.2003.12.029. PMID 15231459
- [Background] Mouzas GL, Yeadon A. Does the choice of suture material affect the incidence of wound infection? A comparison of dexon (polyglycolic acid) sutures with other commonly used sutures in an accident and emergency department. Br J Surg. 1975 Dec;62(12):952-5. doi: 10.1002/bjs.1800621207. PMID 1106807
- [Background] Edwards DJ, Elson RA. Skin closure using nylon and polydioxanone: a comparison of results. J R Coll Surg Edinb. 1995 Oct;40(5):342-3. PMID 8523317
- [Background] Lundblad R, Simensen HV, Wiig JN, Niels Gruner OP. [Skin closure. A prospective randomized study]. Tidsskr Nor Laegeforen. 1989 Apr 30;109(12):1307-9. Norwegian. PMID 2660322
- [Background] Murphy PG, Tadros E, Cross S, Hehir D, Burke PE, Kent P, Sheehan SJ, Colgan MP, Moore DJ, Shanik GD. Skin closure and the incidence of groin wound infection: a prospective study. Ann Vasc Surg. 1995 Sep;9(5):480-2. doi: 10.1007/BF02143863. PMID 8541198
- [Background] Holger JS, Wandersee SC, Hale DB. Cosmetic outcomes of facial lacerations repaired with tissue-adhesive, absorbable, and nonabsorbable sutures. Am J Emerg Med. 2004 Jul;22(4):254-7. doi: 10.1016/j.ajem.2004.02.009. PMID 15258862
- [Background] Luck RP, Flood R, Eyal D, Saludades J, Hayes C, Gaughan J. Cosmetic outcomes of absorbable versus nonabsorbable sutures in pediatric facial lacerations. Pediatr Emerg Care. 2008 Mar;24(3):137-42. doi: 10.1097/PEC.0b013e3181666f87. PMID 18347489
- [Background] Luck R, Tredway T, Gerard J, Eyal D, Krug L, Flood R. Comparison of cosmetic outcomes of absorbable versus nonabsorbable sutures in pediatric facial lacerations. Pediatr Emerg Care. 2013 Jun;29(6):691-5. doi: 10.1097/PEC.0b013e3182948f26. PMID 23714755
- [Background] Tejani C, Sivitz AB, Rosen MD, Nakanishi AK, Flood RG, Clott MA, Saccone PG, Luck RP. A comparison of cosmetic outcomes of lacerations on the extremities and trunk using absorbable versus nonabsorbable sutures. Acad Emerg Med. 2014 Jun;21(6):637-43. doi: 10.1111/acem.12387. PMID 25039547
- [Background] Quinn JV, Drzewiecki AE, Stiell IG, Elmslie TJ. Appearance scales to measure cosmetic outcomes of healed lacerations. Am J Emerg Med. 1995 Mar;13(2):229-31. doi: 10.1016/0735-6757(95)90100-0. PMID 7893315
- [Background] Quinn JV, Wells GA. An assessment of clinical wound evaluation scales. Acad Emerg Med. 1998 Jun;5(6):583-6. doi: 10.1111/j.1553-2712.1998.tb02465.x. PMID 9660284
- [Background] Singer AJ. Clinical wound evaluation scales. Acad Emerg Med. 1998 Jun;5(6):564-6. doi: 10.1111/j.1553-2712.1998.tb02461.x. No abstract available. PMID 9660280